CLINICAL TRIAL: NCT03157102
Title: High Flow Nasal Cannula Versus Standard Oxygen Therapy in Children With Status Asthmaticus: a Randomized Controlled Trial
Brief Title: High Flow Nasal Cannula in Children With Status Asthmaticus
Acronym: CANULASTHM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL17_0035; IDRCB (Other: 2018-A00615-50)
Record Dates: First submitted 2017-05-02; First posted 2017-05-17 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Status Asthmaticus
Keywords: children; status asthmaticus; HFNC
MeSH Terms: conditions — Status Asthmaticus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC group (Experimental)
  Interventions: Device: HFNC
- Standard Oxygen Therapy group (STO group) (Other)
  Interventions: Device: Standard Oxygen Treatment

INTERVENTIONS:
Device: HFNC — Oxygen therapy will be delivered through high flow nasal cannulas. Aerosol treatments will be administered through a vibrating mesh nebulizer directly connected to the circuit (aerogen®). The airvo® system (Fisher & Peykel Healthcare, Auckland, New Zealand) will be used as the high flow cannula system in the study. Cannula size will be tailored to the child according to the manufacturer's recommendations. The gas flow will be adjusted according to the child's weight in a predefined chart. FiO2 will be adjusted to allow for a SpO2 >92%.
  All the patients, regardless of their treatment failure status, will be evaluated at H2, H6, H12 and H24 to monitor their evolution (evaluation of the standard parameters, consciousness, PRAM (Pediatric Respiratory Assessment Measure) score, pain assessment by the FLACC (Face Legs Activity Cry Consolability) score). .
  Arms: HFNC group
Device: Standard Oxygen Treatment — Children will receive supplemental oxygen as commonly delivered through a non-rebreather face mask or low flow nasal cannula (standard oxygen treatment) and beta2 agonist aerosol via vibrating mesh nebulizer (aerogen®) according to the procedures usually used in the unit and according to the GINA (Global Initiative for Asthma) protocol. This group is the standard treatment group and is therefore the control group.
  All the patients, regardless of their treatment failure status, will be evaluated at H2, H6, H12 and H24 to monitor their evolution (evaluation of the standard parameters, consciousness, PRAM score, pain assessment by the FLACC score). The use of adjuvant therapies (magnesium sulfate, salbutamol IVSE, and ipratropium bromide) will remain at the discretion of the physician in charge of the child and will be evaluated as a secondary criterion.
  Arms: Standard Oxygen Therapy group (STO group)

SUMMARY:
In France, over 2.5 million people suffer from asthma, including one-third of children. This is the chronic respiratory disease leading to the highest rate of hospitalization. The conventional oxygen delivery means in children are the non-rebreather face mask or low flow nasal cannula (standard oxygen therapy - SOT). New non-invasive ventilatory support systems such as High Flow Nasal Cannula (HFNC) are emerging. These are nasal cannulas allowing the delivery of a high air (or oxygen) flow, exceeding the inspiratory flow of patients with acute respiratory failure, allowing to deliver a slight positive expiratory pressure while ensuring humidification and warming of the airways. Aerosol administration is also possible with excellent efficiency and without interrupting respiratory assistance. Physiological data and clinical studies in other pathologies suggest the interest of this technique during the asthma attack, but no comparative study currently exists in this indication. The HFNCs could have their place upstream of Non Invasive Ventilation (NIV), thus replacing non-rebreather face mask sometimes not tolerated by the children. The investigators's hypothesis is that HFNCs could improve patients' health faster, reduce the use of other ventilatory assistance (NIV, invasive ventilation) and reduce the duration of hospitalization in intensive care units or continuous monitoring units (CMU).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 6 months and <18 years old
* Hospitalized in PICU with status asthmaticus defined by

  1. a PRAM score > 7 with no response at H2 to the conventional treatment according to the GINA (Global Initiative for Asthma guidelines) protocol: Oxygen therapy, Continuous nebulization of beta2 agonist for at least one hour then every hour, Oral or intravenous corticosteroid (ie methylprednisolone 2mg/kg/j)
  2. or with hypercapnic acidosis (pCO2 > 45 mmHg and pH < 7,35)
* Informed consent signed by at least on parent or legal guardians prior to inclusion and oral consent of the other parent if absent

Exclusion Criteria:

* Non-corrected congenital heart disease, or neuromuscular disease, or chronic respiratory disease (pulmonary or bronchial fibrosis, cystic fibrosis), or ENA disease (laryngo or tracheo malacia), scoliosis or chronic metabolic disease
* Need for non-invasive or invasive ventilation (Glasgow comas scale <8, hemodynamic instability, refractory hypoxemia, cardiac arrest)
* Pneumothorax confirmed on the X-ray
* No national health coverage

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 272 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Number of patients with first line treatment Failure as defined below in the first 24 hours | up to hour 24
  First line treatment Failure in the first 24 hours is defined as:
  * Occurrence or worsening of hypercapnic acidosis (pH<7.35 with pCO2>45 mmHg)
  * Or worsening of PRAM score (>=2 from baseline)
  * Or SpO2<92% with maximal flow of oxygen depending on age in the group standard oxygen therapy or with FiO2 > 60% associated with a flow between 1 and 3L/Kg/min in the HFNC group
  * Or occurrence or worsening of the level of consciousness with Glasgow coma scale < 12
  * Or the need of invasive or noninvasive ventilation (Glasgow coma scale<8, hemodynamic instability, refractory hypoxemia) at any time during the first 24 hours

SECONDARY OUTCOMES:
Number of Patients requiring noninvasive ventilation (NIV) | month 1
Number of Patients requiring invasive ventilation (IV). | month 1
Duration of invasive ventilation (IV). | month 1
  Duration in hours
Duration of noninvasive ventilation (NIV) | month 1
  Duration in hours
Comfort assessed by the FLACC score | up to hour 24
Duration of supplemental oxygen therapy (in hours) | month 1
Time from inclusion to restoration of a PRAM score < 8 (in hours). | month 1
Time from inclusion to blood gas normalization (pCO2<45 mmHg and pH>7.35) if available (hours) | month 1
Cumulative dose of treatments (salbutamol, corticosteroid magnesium sulfate) | month 1
  in milligram during PICU stay
total number of hours of PICU stay | month 1

CONTACTS AND LOCATIONS:
Overall Officials: Robin Pouyau, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (14):
- France (14):
  - Hôpital Femme-Mère-Enfant, Bron
  - CHU de Dijon, Dijon
  - CHU de Grenoble Alpes, Grenoble
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Timone 2, Marseille
  - CH Annecy Genevois, Metz-Tessy
  - CHU Arnaud de Villeneuve, Montpellier
  - CHU de Nantes, Nantes
  - Chu Lenval, Nice
  - Hôpital Armand Trousseau, Paris
  - Hôpital Necker Enfants Malades, Paris
  - Hôpital Robert Debré, Paris
  - CHU Strasbourg,, Strasbourg
  - CH Villefranche sur Saône,, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No